CLINICAL TRIAL: NCT04407624
Title: Effects of Intermittent Exercise Training Programs in Patients With Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Elvan Keles, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4923-GOA
Record Dates: First submitted 2020-01-27; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Myocardial Infarction
Keywords: Aerobic exercise; Intermittent exercise
MeSH Terms: conditions — Myocardial Infarction | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Exercise Group (Experimental): Warm-up, loading (walking, squat, sitting down on a chair, limb movements with weights, stepping on steps, walking on different floors), cooling and relaxation exercises
  Interventions: Other: Intermittent Exercise
- Control Group (Active Comparator): Warm-up, loading (brisk walking at 60-85% of maximum heart rate), cooling and relaxation exercises
  Interventions: Other: Control

INTERVENTIONS:
Other: Intermittent Exercise — Exercise programs including warm-up, loading, cooling, and relaxation exercises are shown. The warm-up period is consist of light-paced walking, active movements of several large muscle groups. During the loading period, taking into consideration the heart rate, fatigue and shortness of breath, exercises such as walking, squat, limb movements with weights, stepping on the steps, walking on different floors are shown. Stretching exercises are done during the cooling period. Intermittent loading workouts will consist of 3-minute loads and 1-minute rest intervals. Participants are contacted every two weeks via communication methods such as e-mail, message and telephone conversation. Exercise diary is given to all patients and is taken from them at the end of the study.
  Arms: Intermittent Exercise Group
Other: Control — Exercise programs including warm-up, loading, cooling, and relaxation exercises are shown. The warm-up period is consist of light-paced walking, active movements of several large muscle groups. In loading period, moderate aerobic exercise is consist of brisk walking to reach 60-85% of the person's maximum heart rate. Stretching exercises are done during the cooling period.
  Arms: Control Group

SUMMARY:
Cardiovascular diseases are a leading cause of death worldwide. According to the World Health Organization (WHO), cardiovascular diseases constitute 1/3 of all causes of death.

Myocardial infarction (MI) is an irreversible myocardial necrosis due to prolonged ischemia.

Patients with MI are candidates for cardiac rehabilitation (CR). American Heart Association (AHA) guidelines recommend exercise-based cardiac rehabilitation and suggest exercise to add to patients' routine treatment. When the literature on patients with MI is examined, various exercise programs are seen. The aims of present study is investigating and comparing the effectiveness of intermittent exercise training and aerobic exercise training programs in patients with MI.

DETAILED DESCRIPTION:
Cases are divided into two groups as exercise (control) and control group by closed envelope randomization method. All patients are informed about risk factors and risk factor management. All patients are trained 3 days in the first week under the supervision of a physiotherapist to learn individual exercise programs. Exercise programs including warm-up, loading, cooling, and relaxation exercises are shown. The warm-up period is consist of light-paced walking, active movements of several large muscle groups. During the loading period, taking into consideration the heart rate, fatigue and shortness of breath, exercises such as walking, squat, limb movements with weights, stepping on the steps, walking on different floors are shown. Stretching exercises are done during the cooling period. Intermittent loading workouts will consist of 3-minute loads and 1-minute rest intervals. Moderate aerobic exercise is consist of brisk walking to reach 60-85% of the person's maximum heart rate. Participants of the experimental group are contacted every two weeks via communication methods such as e-mail, message and telephone conversation. Exercise diary is given to all patients and is taken from them at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Having had MI at least 3 months ago
* Stable clinical status for at least two weeks
* Walking independently
* Volunteer for research study

Exclusion Criteria:

* Having unstable angina
* Having uncontrolled hypertension
* Having hemodynamic instability
* Participating in any exercise program in the last six months
* Having a major orthopedic or neurological problem that limits functionality

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in functional capacity | Baseline, 12th week
  Six-minute walk test (6MWT) is a valid, reliable and useful test for assessing functional capacity of patients. This test assesses distance walked over 6 minutes as a sub maximal test of aerobic capacity/endurance.
Change in peripheral muscle strength | Baseline, 12th week
  The Jamar Handgrip Dynamometer is an instrument for measuring the maximum isometric strength of the hand and forearm muscles.
  Quadriceps isometric muscle strength is measured with a Hand Held Dynamometer.
Change in respiratory muscle strength | Baseline, 12th week
  Measurement of respiratory muscle strength is useful in order to detect respiratory muscle weakness and to quantify its severity. Respiratory muscle strength is assessed by mouth pressures sustained for 1 s during maximal static manoeuvre against a closed shutter.
Change in FEV1 | Baseline, 12th week
  FEV1 is the maximal amount of air which is forcefully exhale in one second. It is then converted to a percentage of normal predicted based on height, weight, and race.
Change in FVC | Baseline, 12th week
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from lungs after taking the deepest breath possible, as measured by spirometry.
Change in FEV1/FVC | Baseline, 12th week
  Also known as Tiffeneau-Pinelli index, FEV1/FVC ratio is often used in diagnosing and treating lung diseases. The FEV1/FVC ratio is a measurement of the amount of air you can forcefully exhale from your lungs.
Change in PEF | Baseline, 12th week
  Peak expiratory flow (PEF) is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration, measured in liters per minute or in liters per second.

SECONDARY OUTCOMES:
Change in weight | Baseline, 12th week
  Tanita Body Composition Analyzer determines body weight as kilograms (kg).
Change in body mass index | Baseline, 12th week
  Tanita Body Composition Analyzer determines Body Mass Index (BMI) which is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Change in body fat percentage | Baseline, 12th week
  Tanita Body Composition Analyzer determines the body fat percentage (BFP) which is the total mass of fat divided by total body mass, multiplied by 100.
Change in lean body mass | Baseline, 12th week
  Tanita Body Composition Analyzer determines Lean Body Mass (LBM) also known as "Fat-Free Mass" which is the total weight of body minus all the weight due to your fat mass. LBM includes the weight of organs, skin, bones, body water and muscle mass.
Change in severity of dyspnoea | Baseline, 12th week
  Modified Medical Research Council (mMRC) dyspnea scale is a valid and reliable test for measuring the severity of dyspnea. This scale ranges from 0 to 4. A higher value represents a worse outcome.
Change in The Tampa Kinesiophobia Scale for Heart Patients | Baseline, 12th week
  The Tampa Kinesiophobia Scale for Heart Patients is a questionnaire consisting of 17 questions evaluating the fear of movement in heart patients. The minimum value is 17 and the maximum value is 68, and the higher score means a worse outcome.
Change in The International Physical Activity Questionnaire-short form | Baseline, 12th week
  The International Physical Activity Questionnaire-short form (IPAQ-SF) consists of 7 questions and gives information about the time spent on walking, moderate-to-severe, severe activities. A score in MET-minutes is obtained. The minimum value is 0 and the higher score means a better outcome.
Change in The Fatigue Severity Scale | Baseline, 12th week
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. The minimum value is 9 and the maximum value is 63. The higher score means greater fatigue severity.
Change in The Hospital Anxiety and Depression Scale | Baseline, 12th week
  The Hospital Anxiety and Depression Scale (HADS) assesses both anxiety and depression, which commonly coexist. It comprises seven questions for anxiety and seven questions for depression, and takes 2-5 min to complete. The minimum value is 0, the maximum value is 21 and the higher score means a worse outcome.
Change in MacNew Heart Disease Health-Related Quality of Life instrument | Baseline, 12th week
  The MacNew Heart Disease Health-related Quality of Life (HRQL) instrument is designed to assess patient's feelings about how ischemic heart disease affects daily functioning and contains 27 items with a global HRQL score and physical limitation and emotional, and social function subscales with a 2-week timeframe. The maximum possible score in any domain is 7 and the minimum is 1. The higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül Üniversitesi School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Yakut H, Dursun H, Felekoglu E, Baskurt AA, Alpaydin AO, Ozalevli S. Effect of home-based high-intensity interval training versus moderate-intensity continuous training in patients with myocardial infarction: a randomized controlled trial. Ir J Med Sci. 2022 Dec;191(6):2539-2548. doi: 10.1007/s11845-021-02867-x. Epub 2022 Jan 7. PMID 34993836
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536